CLINICAL TRIAL: NCT06915012
Title: A Randomized Double-Blinded and Placebo-Controlled Trial to Assess the Impact of Biophoton Therapy on Chronic Severe Arthritis Pain
Brief Title: Impact of Biophoton Therapy on Chronic Severe Arthritis Pain
Acronym: Severe Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Institute of All Medicines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIAM-PN385
Record Dates: First submitted 2025-04-01; First posted 2025-04-07 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-04

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blinded, placebo-controlled intervention clinical study to assess the effectiveness of biophoton therapy in managing chronic severe pain. Approximately 102 patients with chronic severe arthritis pain will participate in the two-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each active or inactive Biophotonizer will be labeled individually with a code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Treatment Arm with Biophoton Therapy (Experimental): This arm is to determine the efficacy of the Biophoton Generator in reducing pain and improving the quality of life of patients with arthritis.
  Interventions: Device: Tesla BioHealing(R) Biophoton Generators
- Comparison Arm treated with Placebo-Device (Placebo Comparator): This arm is to compare with the active devices in reducing pain and improving the quality of life of patients with arthritis.
  Interventions: Device: Tesla BioHealing(R) Biophoton Generators

INTERVENTIONS:
Device: Tesla BioHealing(R) Biophoton Generators — Biophoton generators have been reported to reduce severe chronic pain significantly. This is to determine its efficacy.

SUMMARY:
Study Objective The purpose of this clinical study is to evaluate if biophoton therapy, delivered by Tesla BioHealing® Biophoton Generators (Biophotonizer), can alleviate chronic severe pain.

Study Design This is a randomized, double-blinded, placebo-controlled intervention clinical study to assess the effectiveness of biophoton therapy in managing chronic severe pain. Approximately 102 patients with chronic severe arthritis pain will participate in the study.

Study Randomization The biostatistician will prepare a randomization schedule including a series of subject numbers. A subject number will be randomly assigned to each study participant, which will assign them to either the control group or the treatment group.

Other than the Informed Consent Form (ICF), all study information will be recorded by using the subject number. The Principal Investigator, study physicians, study nurse, data-entry specialists, and biostatisticians, as well as the participants (and caregivers), will be blinded about who received which product during the first two weeks of study participation.

Study Enrollment Each potentially qualified patient will review the Informed Consent Form online (e-ICF) and Enrollment Criteria online (e-Criteria) first, then discuss the e-ICF and e-Criteria with the study team medical professional via telephone during the scheduled time. Each qualified patient will sign the e-ICF and send it to the Study Coordinator. The Study Coordinator will assign the qualified patient a randomized subject number, then the patient will become a study participant.

Study Procedure We expect that the participant will stay in this clinical treatment for 12 weeks, or 12 weeks if the participants are randomly placed in a placebo group. The 12 weeks of participation are double-blinded to record the placebo effects, as each set of the study device is labelled with a unique code for use by only one participant. The change of the placebo device to the treatment device will be performed by the study device management team staff, who will not inform the study participant or study research staff who are involved in study data collection. Each participant assigned to the Control Group will be treated with the 4 placebo devices on the bed. Each participant assigned to the Treatment Group will receive 4 Biophoton generator devices and placed on the bed on each side of the body. Each participant will use the Treatment or Control device for at least 8 hours every night for the 12 weeks during sleep. During the day, participants are welcome to bring the study devices and place them near the bodies during the daytime. At the end of the initial 12 weeks, study participants randomized to the Placebo group will be advised whether they will use the Open-Labeled product to treat them for 4 to 12 weeks. Only the visual analog scale of the pain data will be collected after the switch. Each participant will be guided by study team staff to perform the following tests on their assigned testing days: a visual analog scale, brief pain inventory, pain disability index, the standard SF-36 questionnaires (SF-36) for measuring life quality, the Pittsburgh Sleep Quality Index, a Patient Global Impression of Change, a Hospital Anxiety and Depression Scale, and inflammatory markers that provide objective evidence of inflammation.

Investigational Product and Mode of Administration Tesla BioHealing Biophotonizer is an over-the-counter (OTC) medical device, and it can be used by anyone who wants to increase blood circulation and reduce bodily pains. For this study, the active or inactive Biophotonizer will be labeled with a code. The participant and/or caregiver cannot know if the devices are active or inactive. When the participant places the devices close to the body, she/he may or may not receive life force energy. The participant will record changes in quality of life and complete the standard study questionnaires at baseline and the end of each 2-week interval.

Comparator and Mode of Administration Clinical measurements will be conducted by medical professionals. The same shape, size, and weight of the device without generating biophotons is to be labeled with a random code and used as a comparator. The comparator device will be placed close to the body during sleep during the entire study period. The participant will record the life quality changes and answer the standard study questionnaires. Clinical measurements will be conducted by medical professionals.

Study Duration Estimated date of the first patient enrolled: November 15, 2024. The estimated date of the last patient completed: November 15, 2025.

Participants in the Treatment Group and Control Group will actively participate in the study for 12 or 24 weeks. Each Participant will answer the standard study questionnaires several times, respectively, at the baseline, at the end of each 2-week interval after starting the study treatment.

DETAILED DESCRIPTION:
Outcome Variables

Primary Outcome Measure:

The Visual Analog Scale (VAS) asks participants to rate their arthritis pain on a scale from 0 to 10, and 10 being the worst pain imaginable. [Time Frame: 0-2, 0-4, 0-6, 0-8, 0-10, 0-12 weeks]. VAS has been used worldwide as a standard clinical research tool.

Secondary Outcome Measure:

1. Life Quality. Short Form Health Survey (SF-36) [Time Frame: 0-2, 0-4, 0-6, 0-8, 0-10, 0-12 weeks] is to measure the quality of life as influenced by the investigational medical device. SF-36 has been used worldwide as a standard clinical research tool.
2. Pain Disability Index (PDI) [Time Frame: 0-2, 0-4, 0-6, 0-8, 0-10, 0-12 weeks]. The PDI measures the degree to which pain impacts 7 different categories of daily activities.
3. Hospital Anxiety and Depression Scale (HADS) [Time Frame: 0-2, 0-4, 0-6, 0-8, 0-10, 0-12 weeks]. Chronic pain typically influences anxiety and depression levels, which are measured by HADS.
4. Pittsburgh Sleep Quality Index (PSQI). The PSQI will assess the quality and patterns of sleep in the participants. Chronic pain is often accompanied by changes in sleep quality. [Time Frame: 0-2, 0-4, 0-6, 0-8, 0-10, 0-12 weeks]. This will be verified by using a MUSE EEG to monitor sleeping quality.
5. Inflammatory and Anti-Inflammatory Markers. The laboratory measurement of C-reactive protein (CRP), Tumor Necrosis Factor-alpha (TNF-α), interleukin-6 (IL-6), macrophages, and stem cells provides evidence of changes in inflammation and anti-inflammation related to the pain in the body. This will provide important evidence why biophoton generators can be effective in alleviating chronic severe arthritis pain [Time Frame: baseline, 0-2, 0-4, 0-6, 0-8, 0-10, 0-12 weeks]. The study may allow for cessation of inflammatory and anti-inflammatory marker assessments if a 50% reduction in pain, as measured on the pain scale, is observed.
6. Pain medicine use. The reported pain medicine use will be tabulated and analyzed. [Time Frame: 0-2, 0-4, 0-6, 0-8, 0-10, 0-12 weeks]
7. Neurological Examination by a Study Physician. [Time Frame: 0-2, 0-4, 0-6, 0-8, 0-10, 0-12 weeks].

Safety Outcome: Occurrence of adverse events. Any adverse events were reported by participants. [Time Frame: Any Adverse Events occurred at the baseline, and up to 12 weeks.] Any adverse events reported by participants will be tabulated and compared between the two groups.

Pregnancy Test and Participant Assurance of Non-Pregnancy for Clinical Trial will be given to females of reproductive age/childbearing age. [Time Frame: 0-2, 0-4, 0-6, 0-8, 0-10, 0-12 weeks].

Eligibility Criteria

Inclusion Criteria:

* Willing and able to give informed consent for participation in the trial.
* Is able and willing to comply with all trial requirements.
* Male or female aged 18-80 years old with stable chronic severe pain.
* ≥3 months duration of chronic severe arthritis pain.
* A current VAS pain rating ≥5/10
* Able to complete the treatment for the study period.
* Must be fluent in English.

Exclusion Criteria:

* Untreated psychiatric disturbances that would affect trial participation as judged by the research medical professional.
* Who relies on ventilators
* Co-morbid conditions that would interfere with study activities or response to treatment, which may include severe chronic pulmonary disease, history of uncontrolled seizures, acute or chronic infectious illness, severe diabetes, kidney failure, or any end-of-life prognosis.
* Is participating in another investigational drug or device trial
* Has an active infectious disease, such as COVID-19
* Pregnant women.

Statistical Methods The sample size is calculated based on the primary efficacy variable and the data from the published study in chronic severe arthritis pain (less than 10% success rate) to compare the treatment with the Biophoton Generator, which was at least 50% successful, and to compare with a placebo. The treatment success is defined as a 50% reduction of the visual analog scale at any study week as compared to the baseline. To be conservative, two successful rates, 40%, 50% for the Treatment, 20% for the Control, were used to calculate sample sizes, see table below.

Possibility Number Control Success Rate % Treatment Success Rate* % Power Confidence Level Sample Size per Group Additional 20% per Group 2 20% 50% 90% 95% 19 4

*Treatment success is defined as the pain level reduced by 2/10 VAS at any time during the study.

We plan to enroll 51 Participants in each group to have 42 completers by adding 9 (20%) more participants. Therefore, a total of 102 participants with arthritis pain will be enrolled. If the Principal Investigator decides to increase the enrollment to enable a statistical difference between the two groups with arthritis pain, the enrollment can be continued. Primary and secondary outcome variables will be statistically analyzed by using Chi-square analysis or paired T-Test.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the trial.
* Is able and willing to comply with all trial requirements.
* Male or female aged 18-80 years old with chronic severe arthritis pain.
* ≥3 months duration of chronic severe arthritis pain.
* a current VAS pain rating ≥5/10.
* Able to complete the treatment for the study period.
* Must be fluent in English.

Exclusion Criteria:

* Untreated psychiatric disturbances that would affect trial participation as judged by the Caregiver or by the clinical study medical professional
* Who relies on ventilators
* Who had deep brain stimulators, or pacemakers, or implantable electronic devices
* Co-morbid conditions that would interfere with study activities or response to treatment, which may include severe chronic pulmonary disease, history of uncontrolled seizures, acute or chronic infectious illness, severe diabetes, kidney failure, or any end-of-life prognosis.
* Is participating in another investigational drug or device trial
* Has an active infectious disease, such as COVID-19
* Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
To determine if treatment with Biophoton Generator can significantly reduce arthritis pain | 3 months
  VAS score to measure reduction in pain levels

SECONDARY OUTCOMES:
To determine if treatment with Biophoton Generator can significantly improve life quality | 3 months
  Quality of life Questionnaires Summarized as SF-36 Score
If the use of pain killer can be reduced | 3 months
  Study questionnaire of pain killer use

CONTACTS AND LOCATIONS:
Overall Officials: James Z Liu, MD, PhD, Study Chair — First Institute of All Medicines
Locations (1):
- Tesla BioHealing Medical Center in Butler-PA, Butler, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) might not be shared due to concerns regarding participant privacy, confidentiality, and compliance with ethical and regulatory guidelines. Additionally, data sharing may be restricted by the terms of informed consent or institutional review board (IRB) approval.

REFERENCES:
- See also: Related Info — https://doi.org/10.1080/14653240600855905